CLINICAL TRIAL: NCT05211596
Title: Deaf Weight Wise: Community-engaged Implementation Research to Promote Healthy Lifestyle Change With Deaf American Sign Language Users in Western and Central New York State
Brief Title: Deaf Weight Wise: Community-engaged Implementation Research to Promote Healthy Lifestyle Change With Deaf ASL Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Steve Barnett, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005784
Record Dates: First submitted 2021-12-25; First posted 2022-01-27 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Healthy Lifestyle; Overweight; Obesity; Cardiovascular Risks; Implementation Research
Keywords: Deaf; American Sign Language
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Intervention Arm (Main Intervention) (Other): Main Intervention
  Interventions: Behavioral: Deaf Weight Wise intervention

INTERVENTIONS:
Behavioral: Deaf Weight Wise intervention — The DWW intervention consists of groups of 5 subjects who meet together for 16 weeks, 2 hours each week. Group meetings will be held virtually on Zoom. A trained, deaf, ASL-fluent counselor will lead the sessions. Each session includes group sharing, problem solving, discussion of a weight management topic, and goal setting and action planning for the next week. A key principle of DWW is motivational interviewing, in which the counselor acts as a facilitator to help participants identify/recognize their own unhealthy behaviors, help individuals build skills that will promote behavior change, and help group members to support each other to make behavior changes. The maintenance phase starts immediately after the 16-week intervention, and consists of two meetings of the original group via Zoom; one at month 3 and one at month 6 of the maintenance period. Counselors also email participants bi-weekly to check in and provide additional support.
  Other Names: DWW

SUMMARY:
The purpose of the Deaf Weight Wise Implementation Study is to study with diverse partners the approaches and strategies that lead to successful implementation of Deaf Weight Wise (DWW), an evidence-based healthy lifestyle intervention for use with Deaf adult American Sign Language (ASL) users. The implementation hypothesis is that diverse community organizations will successfully implement DWW with their constituents.

DETAILED DESCRIPTION:
Little is known about health or health promoting interventions in Deaf communities nationally or worldwide. Deaf individuals comprise understudied and medically underserved populations. Access to health services, research, and health information is confounded by communication and literacy barriers. One of the challenges of health research with deaf people is creating survey instruments and interventions that are culturally and linguistically appropriate. The original Deaf Weight-Wise Study (2012-2014) by this study team of the Rochester Prevention Research Center (RPRC): National Center for Deaf Health Research (NCDHR) was the first adequately powered randomized trial of an evidence-based healthy weight/lifestyle intervention to be carried out in Deaf people. Deaf Weight Wise is based on the University of North Carolina's Weight Wise program and represented a pioneering effort to collect new health information and develop intervention tools in a very understudied and underserved minority group. Deaf Weight Wise 2.0 (2017-2019) was built on this research team's experience with the original Deaf Weight Wise trial for ages 40-70, and was an adaptation of the original Deaf Weight Wise curriculum to suit ages 21-70. DWW 2.0 also evaluated the additional component of a one-to-one individual counseling intervention delivered remotely over videophone (like Skype/Zoom) in addition to the group intervention format.

This new Deaf Weight Wise implementation research proposed here will allow this study team to work with community partner organizations, to train them to implement DWW at their own sites. This will fulfill the goal of disseminating DWW broadly to Deaf communities. The study team will conduct research to study the process of implementation of DWW at each site. This advances DWW along the translational spectrum to ensure that DWW is not only a research project, but becomes a sustainable, community-based program.

The study team will conduct an implementation-effectiveness Type 3 research design that is plan, execute and evaluate in collaboration with partners. The study team will adapt and implement DWW with partner organizations at various sites in central and western NY. Each phase of this study, including selection of the intervention topic (obesity and healthy lifestyle), design of study procedures, and development of the informed consent and data collection processes, are based on direct input and feedback from Deaf research team members and Deaf community members.

All aspects of this research will be conducted via virtual video communication platforms.

Screening and enrollment is conducted in American Sign Language by Deaf sign-fluent research staff. Informed consent is an ASL video followed by discussion, question and answer, and check for comprehension in ASL by Deaf sign-fluent research staff. Following informed consent, subjects will have data collection appointments at baseline (pre-intervention), 6-months after baseline (post-intervention), and 18-months after baseline (1 year post-intervention). Data collection surveys are conducted via online ASL video surveys with English text support. Data collection interviews at all data collection points are conducted by Deaf sign-fluent research staff.

Following baseline appointments, a trained Deaf sign-fluent DWW intervention counselor from each implementation site will lead the group intervention via virtual video communication platform, with about 5 participants per group. As additional participants are enrolled, new groups will be formed (rolling enrollment at each site).

ELIGIBILITY:
Inclusion Criteria:

• Deaf people who use sign language and live in one of the following three regions: Buffalo NY, Rochester NY, or Syracuse NY and/or part of the typical clientele/populations that the implementation partner sites serve;

AND:

* Are Ages 18 and older
* Have a body mass index (BMI) of 18.5 or higher (normal BMI category or higher).
* Eligible subjects who wish to participate in the intervention component of the program (16-weeks plus 6-month maintenance phases) must also have permission from a healthcare provider to participate in the intervention if: 1) self-reported diagnosis of a recent cardiovascular disease event (heart attack or stroke in past 6 months), 2) self-reported heart condition, chest pain, dizziness, or other reason not to participate in physical activity, 3) had weight loss surgery in the previous 2 years (self-reported), 4) are pregnant (self-reported), and 5) has a BMI over 45.
* Subjects must also be willing to follow a healthy dietary pattern and to abstain from using weight loss medications during the study, and be willing and able to attend group sessions, and to participate in data collection requirements.

Exclusion Criteria:

* Those who are unable or unwilling to provide informed consent, and are unable to see and interact with computer-based questionnaires and educational interventions.
* Subjects with any of the following conditions who wish to participate in the intervention component of the program but do not have permission from a clinician may be instructed to abstain from specific intervention components, including those who reported 1) a cardiovascular disease event in the past six months, 2) or heart condition, chest pain, dizziness, or other reason not to participate in physical activity, 3) or weight loss surgery in the past two years, 4) are pregnant, or 5) has a BMI over 45.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Barnett, MD, Principal Investigator — University of Rochester
Locations (1):
- National Center for Deaf Health Research, University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of this study, deidentified participant dataset may be made available to interested researchers who fully complete the NCDHR Data Use agreement Process. This process includes a requirement to present the research plan to the NCDHR Research Committee and relevant Community Committee no more than 90 days prior to beginning the research project. In addition, results must be presented to the NCDHR Research Committee and relevant Community Committee within a 60-day period following the completion of the research project.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After completion of this study.
Access Criteria: Access to deidentified data will only be granted if the interested researcher fully completes the NCDHR Data Use agreement Process.

REFERENCES:
- [Background] Samuel-Hodge CD, Johnston LF, Gizlice Z, Garcia BA, Lindsley SC, Bramble KP, Hardy TE, Ammerman AS, Poindexter PA, Will JC, Keyserling TC. Randomized trial of a behavioral weight loss intervention for low-income women: the Weight Wise Program. Obesity (Silver Spring). 2009 Oct;17(10):1891-9. doi: 10.1038/oby.2009.128. Epub 2009 Apr 30. PMID 19407810
- [Background] Barnett S, Matthews K, DeWindt L, Sutter E, Samuel-Hodge C, Yang H, Pearson TA; Deaf Weight Wise Study Group. Deaf Weight Wise: A novel randomized clinical trial with Deaf sign language users. Obesity (Silver Spring). 2023 Apr;31(4):965-976. doi: 10.1002/oby.23702. Epub 2023 Mar 8. PMID 36890106
- See also: NCDHR Deaf Weight Wise research website — https://www.urmc.rochester.edu/ncdhr/research/current-research/deaf-weight-wise-western-ny.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through various methods (e.g., outreach at community sites, social media) and enrolled on a rolling basis. The first participant was enrolled on Feb. 2, 2022, and the last on Aug. 1, 2023.
Pre-assignment Details: All participants who completed the baseline survey and provided consent were considered enrolled.
Groups:
- Behavioral: Deaf Weight Wise Intervention: Deaf Weight Wise is a group intervention lead by trained, American Sign Language (ASL)-fluent coaches, who utilize an existing evidence-based curriculum that emphasizes healthy eating, exercise, and lifestyle components. It is a behavior change intervention that uses motivational interviewing techniques to help participants identify/recognize unhealthy behaviors, build skills that will promote behavior change, and help group members to support each other to make behavior changes.
  Following baseline appointments, a coach from each implementation site led the group intervention via virtual video communication platform (Zoom), with about 5 participants per group. As additional participants enrolled, new groups were formed. Subjects were asked to complete a daily food and physical activity diary during the 16-week curriculum. Each session included a weigh-in, personal sharing and problem solving, discussion of a weight management topic, and a discussion on goal setting and action planning for the next week. After the 16-week curriculum, the intervention included a 6-month follow up and an 12-month maintenance phase.
  Following informed consent, data collection surveys were conducted via online ASL video surveys with English text support at baseline (pre-intervention), 6 months after baseline (post-intervention), and 18 months after baseline (post-maintenance). Data collection interviews at all data collection points were conducted by ASL-fluent research staff.
Period: Baseline to 6 Months
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Started | 85
Completed | 72
Not Completed | 13
Not completed — Lost to Follow-up | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Period: 6 Months to 18 Months
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Started | 72
Completed | 63
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.66 (13.76)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 60
  Male | 22
  Other | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 62
  More than one race | 5
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: Participants] — Study locations were all in Western New York (i.e., Buffalo, Rochester, or Syracuse)
  Participants
    United States | 85
Age Became Deaf [Count of Participants; unit: Participants] — Self-reported age at which participant became deaf
  Participants
    Became deaf at age 3 or younger (incl. born deaf) | 73
    Became deaf at age 4 or older | 4
    Unknown | 7
    Not reported | 1
Number of participants enrolled at each Implementation Site [Count of Participants; unit: Participants] — Nine partner sites in Western NY initially agreed to provide Deaf Weight Wise (DWW). Two in Buffalo (BUF), five in Rochester (ROC), two in Syracuse (SYR). In addition, 5 participants are not included in this baseline measure because they were not recruited through a site, they were recruited directly online with NCDHR. Population: 5 participants are not included in this baseline measure because they were not recruited through a site, they were recruited directly online with NCDHR.
  Participants
    Rochester View Apartments (ROC): number analyzed (Participants) | 80
    Rochester View Apartments (ROC) | 11
    Deaf Wellness Center (ROC): number analyzed (Participants) | 80
    Deaf Wellness Center (ROC) | 11
    Rochester Institute of Technology (ROC): number analyzed (Participants) | 80
    Rochester Institute of Technology (ROC) | 23
    Rochester Recreation Club for the Deaf (ROC): number analyzed (Participants) | 80
    Rochester Recreation Club for the Deaf (ROC) | 13
    YMCA of Greater Rochester (ROC): number analyzed (Participants) | 80
    YMCA of Greater Rochester (ROC) | 4
    Deaf Access Services (of People, Inc.) (BUF): number analyzed (Participants) | 80
    Deaf Access Services (of People, Inc.) (BUF) | 5
    Buffalo Club for the Deaf (BUF): number analyzed (Participants) | 80
    Buffalo Club for the Deaf (BUF) | 0
    WHOLE ME, Inc. (SYR): number analyzed (Participants) | 80
    WHOLE ME, Inc. (SYR) | 13
    Aurora of Central, NY (SYR): number analyzed (Participants) | 80
    Aurora of Central, NY (SYR) | 0

OUTCOME MEASURES:

1. Primary Outcome: Implementation of the Deaf Weight Wise Intervention at Partner Sites
Description: This outcome measures implementation of the Deaf Weight Wise (DWW) intervention at partner sites, defined as the number of sites that enrolled participants.
Time Frame: Baseline to 18 Months
Measure: Count of Units; unit: Partner Sites
Units Other Than Participants: Partner Sites
Groups:
- Deaf Weight Wise Intervention Partner Site Implementation: The DWW study team worked with community partner organizations to train them to implement DWW at their own sites. The goal was to disseminate DWW broadly to Deaf communities. Working with partner organizations, the study team adapted DWW and supported implementation at various sites in central and western NY. The study team conducted an implementation-effectiveness Type 3 research design to plan, execute, and evaluate in collaboration with partners. Through the process, the study team evaluated whether DWW was implemented and whether it was delivered as intended.
Arm/Group | Deaf Weight Wise Intervention Partner Site Implementation
Number analyzed (Participants) | 80
Number analyzed (Partner Sites) | 9
Partner Sites | 7

2. Primary Outcome: Delivery of the Deaf Weight Wise Intervention As Intended
Description: This outcome measures the number of partner sites that delivered the Deaf Weight Wise (DWW) intervention as intended, based on predefined fidelity criteria (e.g., delivery by site-based coaches, completion of all planned sessions, adherence to the DWW curriculum). Fidelity was assessed through direct observation of sessions and bi-weekly counselor meetings. All intervention sessions were delivered remotely by NCDHR coaches via Zoom.
Time Frame: Baseline to 18 Months
Measure: Count of Units; unit: Partner Sites
Units Other Than Participants: Partner Sites
Arm/Group | Deaf Weight Wise Intervention Partner Site Implementation
Number analyzed (Participants) | 80
Number analyzed (Partner Sites) | 9
Partner Sites | 0

3. Primary Outcome: Number of Participants Who Did Not Receive the Intervention at Their Partner Site Because of Site Barriers and/or COVID Restrictions
Time Frame: baseline to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 85
Participants | 85

4. Secondary Outcome: Participant-Level Outcome: Mean Difference From Baseline to 6 Months (Pre- to Post-Intervention) in Number of Fruit and Vegetable Servings Per Day as Measured by the Block Fruit-Vegetable-Fiber Screener
Description: The mean difference from baseline to 6 months (pre- to post-intervention) in self-reported fruit and vegetable servings per day as measured by the Block Fruit-Vegetable-Fiber Screener.
  The Block Fruit-Vegetable-Fiber Screener is a 10-question survey with responses ranging from: (1) Less than 1/week to (5) 2+/day for each question. An algorithm is then used that incorporates the respondent's age and sex with the additive score from the questions to calculate the Predicted Value for Fruit and Vegetable Servings (Per Day).
Time Frame: Baseline to 6 Months (Pre- to Post-Intervention)
Population: Data from 67 participants were used in this analysis. Of the 72 participants who completed the first period of the intervention (baseline to 6 months), 5 did not submit the Block Fruit-Vegetable-Fiber Screener.
Measure: Mean (Standard Deviation); unit: Fruit and Vegetable Servings per Day
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 67
Fruit and Vegetable Servings per Day
  Baseline | 5.70 (1.56)
  6 Months | 6.13 (1.55)
Statistical Analysis 1: Comparison: Behavioral: Deaf Weight Wise Intervention; Test type: Superiority; p = 0.008, t-test, 2 sided; Mean Difference (Net) = 0.43

5. Secondary Outcome: Participant-Level Outcome: Mean Difference From Baseline to 18 Months (Pre-Intervention to Post-Maintenance) in Number of Fruit and Vegetable Servings Per Day as Measured by the Block Fruit-Vegetable-Fiber Screener
Description: The mean change from baseline to 18 months in self-reported physical activity as measured by the International Physical Activity Questionnaire (IPAQ) - Short Form. The IPAQ records days/week and minutes/day of walking, moderate, and vigorous activity. Scores are expressed in MET-minutes/week using standard values (Walking = 3.3, Moderate = 4.0, Vigorous = 8.0). The total IPAQ score is the sum of all activity categories. Scale range: minimum = 0 (no activity); no fixed maximum, values increase with more activity. Higher scores = better outcome (greater physical activity).
Time Frame: Baseline to 18 Months (Pre-Intervention to Post-Maintenance)
Population: Data from 58 participants were used in this analysis. Of the 63 participants who completed the second period of the intervention (baseline to 18 months), 5 did not submit the Block Fruit-Vegetable-Fiber Screener.
Measure: Mean (Standard Deviation); unit: Fruit and Vegetable Servings per Day
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 58
Fruit and Vegetable Servings per Day
  Baseline | 5.62 (1.57)
  18 Months | 5.83 (1.32)
Statistical Analysis 1: Comparison: Behavioral: Deaf Weight Wise Intervention; Test type: Superiority; p = 0.264, t-test, 2 sided; Mean Difference (Net) = 0.22

6. Secondary Outcome: Participant-Level Outcome: Mean Difference From Baseline to 6 Months (Pre-Intervention to Post-Intervention) in Physical Activity as Reported on the International Physical Activity Question (IPAQ)
Description: The mean change from baseline to 6 months in self-reported physical activity as measured by the International Physical Activity Questionnaire (IPAQ) - Short Form. The IPAQ records days/week and minutes/day of walking, moderate, and vigorous activity. Scores are expressed in MET-minutes/week using standard values (Walking = 3.3, Moderate = 4.0, Vigorous = 8.0). The total IPAQ score is the sum of all activity categories. Scale range: minimum = 0 (no activity); no fixed maximum, values increase with more activity. Higher scores = better outcome (greater physical activity).
Time Frame: Baseline to 6 Months (Pre- to Post-Intervention)
Population: Data from 57 participants were used in this analysis. Of the 72 participants who completed the first period of the intervention (baseline to 6 months), 15 did not submit the 6-month IPAQ.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 57
Score on a scale
  Baseline | 1611.43 (1588.29)
  6 Months | 2460.79 (1965.77)
Statistical Analysis 1: Comparison: Behavioral: Deaf Weight Wise Intervention; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Net) = 849.35

7. Secondary Outcome: Participant-Level Outcome: Mean Difference From Baseline to 18 Months (Pre-Intervention to Post-Maintenance) in Physical Activity as Reported on the International Physical Activity Question (IPAQ)
Description: The mean difference from baseline to 18 months (pre-intervention to post-maintenance) in self-reported physical activity levels over the past 7 days as reported on the International Physical Activity Question (IPAQ).
Time Frame: Baseline to 18 Months (Pre-Intervention to Post-Maintenance)
Population: Data from 50 participants were used in this analysis. Of the 63 participants who completed the second period of the intervention (baseline to 18 months), 13 did not submit the 18-month IPAQ.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 50
Score on a scale
  Baseline | 1409.73 (1481.73)
  18 Months | 2187.14 (2527.10)
Statistical Analysis 1: Comparison: Behavioral: Deaf Weight Wise Intervention; Test type: Superiority; p = 0.054, t-test, 2 sided; Mean Difference (Net) = 777.42

8. Secondary Outcome: Participant-Level Outcome: Mean Percentage Difference From Baseline to 6 Months (Pre- to Post-Intervention) in Self-Reported Body Weight, for Participants With BMI Above Normal Range
Description: The mean weight difference from baseline to 6 months (pre- to post-intervention), expressed as a percentage of baseline weight (in kg), for any participants with a BMI above 24.9 (above normal range)
Time Frame: Baseline to 6 Months (Pre- to Post-Intervention)
Population: Data from 63 participants were used in this analysis. Out of 76 participants with a BMI > 24.9, 63 had weight data at 6 months.
Measure: Mean (Standard Deviation); unit: percentage of baseline weight
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 63
percentage of baseline weight
  Baseline | 0.00 (0.00)
  6 Months | -0.04 (0.05)
Statistical Analysis 1: Comparison: Behavioral: Deaf Weight Wise Intervention; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.04

9. Secondary Outcome: Participant-Level Outcome: Mean Percentage Difference From Baseline to 18 Months (Pre-Intervention to Post-Maintenance) in Self-Reported Body Weight, for Participants With BMI Above Normal Range
Description: The mean weight difference from baseline to 18 months (pre-intervention to post-maintenance), expressed as a percentage of baseline weight (in kg), for any participants with a BMI above 24.9 (above normal range)
Time Frame: Baseline to 18 Months (Pre-Intervention to Post-Maintenance)
Population: Data from 56 participants were used in this analysis. Out of 76 participants with a BMI > 24.9, 56 had weight data at 18 months.
Measure: Mean (Standard Deviation); unit: percentage of baseline weight
Arm/Group | Behavioral: Deaf Weight Wise Intervention
Number analyzed (Participants) | 56
percentage of baseline weight
  Baseline | 0.00 (0.00)
  18 Months | -0.04 (0.06)
Statistical Analysis 1: Comparison: Behavioral: Deaf Weight Wise Intervention; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Net) = 0.04

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Behavioral: Deaf Weight Wise Intervention
All-Cause Mortality (participants affected / at risk) | 1/85
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT05211596/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT05211596/ICF_001.pdf